CLINICAL TRIAL: NCT06806059
Title: Prospective Randomized Interventional Study to Investigate the Impact of Preoperative Physical Activity on Perioperative Morbidity Following Radical Cystectomy
Brief Title: Preoperative Physical Activity Before Radical Cystectomy and the Impact on Morbidity
Acronym: PRACTICE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Yannic Volz, Principal investigator, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 24-0096
Record Dates: First submitted 2025-01-15; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Urothelial Carcinoma Bladder
Keywords: physical activity; preoperative; cystectomy; activity tracker; physical fitness; complication
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physical Activity (Experimental): The intervention group will engage in increased physical activity, aiming for a daily step count of at least 8,000, with a target of 10,000 steps, over a four-week preoperative period. Weekly supervised phone consultations will be conducted to provide guidance and support.
  Interventions: Behavioral: Physical Activity
- Controll (No Intervention): The control group will track their daily physical activity without being required to meet a specific step target. Weekly phone consultations will still be conducted to monitor and support the participants.

INTERVENTIONS:
Behavioral: Physical Activity — The intervention group will engage in increased physical activity, aiming for a daily step count of at least 8,000, with a target of 10,000 steps, over a four-week preoperative period. Weekly supervised phone consultations will be conducted to provide guidance and support.
  Arms: Physical Activity

SUMMARY:
Bladder cancer (BC) is the 6th most common tumor in Europe, with over 540,000 new cases globally each year. While 75% of cases are non-muscle-invasive and treated bladder-preservingly, muscle-invasive, non-metastatic BC requires radical cystectomy (RC), often with neoadjuvant chemotherapy. RC has one of the highest complication rates in urology, and rehabilitation focuses on mitigating functional impairments, restoring physical and mental capacity, and enabling a swift return to daily life.

The ERAS (Enhanced Recovery After Surgery) protocol has shown benefits in reducing hospital stays without increasing complications in RC. Prehabilitation studies in cancer patients have demonstrated improvements in strength and fitness, though without significant reductions in complications or mortality.

This prospective randomized study, conducted over three years at the University of Munich, will evaluate the effect of preoperative physical activity on perioperative morbidity (primary endpoint). Secondary endpoints include quality of life, hospital stay, mortality, and postoperative physical activity. The intervention group will target 8,000-10,000 daily steps for four weeks preoperatively, monitored via pedometers. Follow-ups will assess physical activity and quality of life at specific intervals pre- and post-surgery.

DETAILED DESCRIPTION:
In Europe, bladder cancer (BC) is the 6th most common tumor entity. Globally, over 540,000 new cases have been reported annually in recent years. Approximately 75% of cases are diagnosed as non-muscle-invasive BC at initial presentation, which can generally be treated in a bladder-preserving manner through transurethral resection and intravesical therapy. In cases of muscle-invasive, non-metastatic BC, guidelines recommend radical cystectomy (RC) with neoadjuvant chemotherapy in a curative setting, provided the patient is suitable for such treatment. Considering comorbidities, mortality, and quality of life, various forms of urinary diversion are employed during RC. These include incontinent diversions, such as ileal or colonic conduits, and continent diversions, such as orthotopic bladder replacement using the ileum (neobladder).

A direct comparison of these different urinary diversion methods is currently challenging due to a lack of data. RC is associated with one of the highest complication rates among urological procedures. Rehabilitation following RC must focus on addressing postoperative functional impairments, restoring physical and mental performance, and facilitating a prompt return to social and professional life. The ERAS (Enhanced Recovery After Surgery) concept, originally established in colorectal surgery, has also demonstrated reduced overall hospital stays in RC without increasing complication rates. While it remains uncertain whether the ERAS concept improves prognosis and morbidity, it is considered safe, as no studies have reported an increase in severe complications or mortality associated with its implementation.

Studies in visceral surgery involving prehabilitation for patients with colorectal, esophageal, and lung cancers have shown functional benefits, such as improved fitness, mobility, and strength, but without reductions in complication rates or mortality. In a randomized controlled trial, Minella EM et al. demonstrated the effectiveness of prehabilitation in improving functional outcomes, such as strength and endurance, in BC patients undergoing RC. However, no significant differences in postoperative complications or mortality were observed. A recent prospective study involving patients prior to RC also reported significant improvements in strength and functional fitness.

In the prospective randomized study presented here for evaluation, the investigators aim to investigate the impact of preoperative physical activity on perioperative morbidity (primary endpoint). Secondary endpoints include quality of life, length of hospital stay, mortality, and postoperative physical activity. The intervention group will undergo preoperative preparation over four weeks, targeting a daily step count of 8,000-10,000. Step counts will be self-monitored by patients using pedometers. Physical activity and quality of life will be assessed at specific time points using established fitness assessments and questionnaires. Comparative follow-ups will take place four weeks before surgery, the day before surgery, one week postoperatively, and at three and twelve months postoperatively.

The study will be conducted as a single-center trial at the Department of Urology at the University of Munich over a three-year period.

ELIGIBILITY:
Inclusion Criteria:

* Urothelial cell cancer of the bladder
* Treatment with radical cystectomy

Exclusion Criteria:

* Need for walking aid
* Depression
* cardiovascular, neuromuscular or orthopaedic deficites / disorders
* Time to surgery < 3 Weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2024-11-29 (Actual); Primary Completion 2026-11-29 (Estimated); Study Completion 2027-11-29 (Estimated)

PRIMARY OUTCOMES:
Perioperative Complications | From surgery to 90 days postoperatively
  Complications that occur during the postoperative hospital stay

SECONDARY OUTCOMES:
Physical Fitness Gripstrength | From the day before the surgery as well as up to 12 months after the surgery
  Kg
HRQOL EORTC-QLQC30 | postoperatively, 3 months and 12 months
  Score indicating quality of life in different subscales: symptoms and functioning scores. Scores reach from 0 to 100. 0 indicating no symptoms in the respective scale, 100 representing a strong symptom. For functioning scores 100 indicate a good functioning, 0 indicate no functioning.
Patients in need for analgesia | From the day before the surgery up to the discharge from the hospital up to 12 months
  The type of medication as well as dosage and times the patient need the medication.
6 Minute Walking Test | During the hospitalisation period until 12 months postoperatively
  Walking distance in meters in 6 minutes
Patients in need of laxatives | From the day before the surgery up to the discharge from the Hospital up to 12 months
  The type of laxative as well as dosage and times the medication is needed

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, LMU Hospital, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No
Ethical and legal obligations